CLINICAL TRIAL: NCT05492708
Title: Children's Health in the Heartland Study
Brief Title: The Heartland Study
Status: Recruiting | Type: Observational
Sponsor: Heartland Health Research Alliance (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: HHRA-HS-Phase1-2019
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy Related; Pregnancy Complications; Birth Defect; Gestational Age and Weight Conditions; Spontaneous Abortion; Miscarriage; Exposure to Herbicides
Keywords: pesticide exposure; birth outcomes; biomonitoring
MeSH Terms: conditions — Pregnancy Complications; Congenital Abnormalities; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal and paternal urine samples, and maternal, paternal, and infant buccal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Heartland Study is a prospective, observational study that will enroll up to 2,600 pregnant participants across the Heartland States in the U.S..

The objective of the Heartland Study is to address major knowledge gaps concerning the health effects of herbicides on maternal and infant health. The study is being conducted to evaluate the associations between environmental exposures to herbicides during and after pregnancy and reproductive health outcomes. The study is measuring multiple biomarkers of herbicide exposure among pregnant Midwesterners and their partners to evaluate associations with pregnancy and childbirth outcomes, epigenetic biomarkers of exposure, and child development.

DETAILED DESCRIPTION:
During Phase 1 of the Study, newly pregnant mothers will be enrolled less than or equal to 20 weeks + 6 days gestation and followed through to the end of pregnancy. Prenatal urine and buccal (cheek) samples will be collected to measure urinary herbicide exposure levels and to identify herbicide induced epigenetic biomarkers. Pregnancy outcomes and fetal health will be documented and analyzed to further investigate potential effects of fetal exposure. Indirect measures such as food and beverage consumption, workplace and household related chemical exposures, substance use, residential proximity to agricultural fields, and socioeconomic factors will be captured from questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant persons ages 18 or older at time of consent who are ≤20+6 weeks pregnant. Best clinical estimate of gestational age will be utilized for recruitment purposes. Enrollment in the first trimester (≤ 13 + 6) is preferred, but anyone ≤ 20 +6 is permitted.
* Living in one of the 13 Heartland Study region states at the time of enrollment (Arkansas, Illinois, Indiana, Iowa, Kansas, Michigan, Minnesota, Missouri, Nebraska, North Dakota, Ohio, South Dakota, or Wisconsin) Optional inclusion of the putative biological father

Exclusion Criteria:

* Participants who are not fluent in and/or do not fully understand, read, write, or speak the English language.
* Other inability to provide informed consent to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants must live in one of the 13 Heartland states at the time of enrollment: Arkansas, Illinois, Indiana, Iowa, Kansas, Michigan, Minnesota, Missouri, Nebraska, North Dakota, Ohio, South Dakota, Wisconsin.
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2020-01-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Pregnancy loss | Enrollment to birth
  Number of participants who experience a pregnancy loss
Preterm birth | Enrollment to gestational age 36 +6
  Number of births that occur between gestational age 20 +0 and 36 +6
Hypertensive disorders of pregnancy | Enrollment to up to twelve weeks after delivery
  Number of participants diagnosed with a hypertensive disorder of pregnancy

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Iowa Health Care, Iowa City, Iowa
  - Gundersen Health, La Crosse, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parvez S, Gerona RR, Proctor C, Friesen M, Ashby JL, Reiter JL, Lui Z, Winchester PD. Glyphosate exposure in pregnancy and shortened gestational length: a prospective Indiana birth cohort study. Environ Health. 2018 Mar 9;17(1):23. doi: 10.1186/s12940-018-0367-0. PMID 29519238
- [Derived] Freisthler M, Winchester PW, Young HA, Haas DM. Perinatal health effects of herbicides exposures in the United States: the Heartland Study, a Midwestern birth cohort study. BMC Public Health. 2023 Nov 22;23(1):2308. doi: 10.1186/s12889-023-17171-9. PMID 37993831
- See also: Sponsor Website — http://hh-ra.org
- See also: Study Webpage — http://hh-ra.org/the-heartland-study